CLINICAL TRIAL: NCT06413563
Title: Analysis of Peripheral Blood Lymphocytes in Patients With Juvenile Idiopathic Arthritis With Respect to Disease Subtypes and Therapy
Status: Not yet recruiting | Type: Observational
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Hager Ibrahim Abdelaal, assisstant lecturer in physical medicine,rheumatology and erhabilitation- sohag university, Sohag University
Other Study IDs: soh-Med-24-04-03MD
Record Dates: First submitted 2024-05-09; First posted 2024-05-14 (Actual); Last update posted 2024-05-14 (Actual); Status verified 2024-05

CONDITIONS: Juvenile Idiopathic Arthritis
MeSH Terms: conditions — Arthritis, Juvenile | interventions — Blood Cell Count

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- juvenile idiopathic arthritis: Juvenile idiopathic arthritis (JIA) is the most common chronic rheumatic disease in children JIA is an umbrella term defining several forms of chronic arthritis with an onset before the age of 16 years, persisting for more than six weeks and with an unknown cause.
  Based on the current International League of Associations in Rheumatology classification criteria (ILAR 2003) , different subtypes of JIA can be distinguished, essentially by a very limited set of clinical features (number of affected joints in the first six months of disease, extra-articular manifestations like fever or features of psoriasis) and serology (presence or absence of rheumatoid factor, RF). The most frequently diagnosed JIA subtypes are oligoarticular JIA (oJIA), polyarticular JIA (pJIA), and systemic JIA (sJIA). Less frequently occurring subtypes are enthesitis-related JIA, psoriatic arthritis, and undefined arthritis. complete blood count will be done for all patients
  Interventions: Diagnostic Test: Complete blood count
- control group: control
  Interventions: Diagnostic Test: Complete blood count

INTERVENTIONS:
Diagnostic Test: Complete blood count — Complete blood count will be done for all patients and then will search about CD4, CD8 T lymphocyte cells surface markers
  * CD56 Natural killer cells surface marker
  * CD19 Lymphocyte cells surface marker

SUMMARY:
Juvenile idiopathic arthritis (JIA) is the most common chronic rheumatic disease in children.

JIA is an umbrella term defining several forms of chronic arthritis with an onset before the age of 16 years, persisting for more than six weeks and with an unknown cause.

Based on the current International League of Associations in Rheumatology classification criteria (ILAR 2003) , different subtypes of JIA can be distinguished, essentially by a very limited set of clinical features (number of affected joints in the first six months of disease, extra-articular manifestations like fever or features of psoriasis) and serology (presence or absence of rheumatoid factor, RF). The most frequently diagnosed JIA subtypes are oligoarticular JIA (oJIA), polyarticular JIA (pJIA), and systemic JIA (sJIA). Less frequently occurring subtypes are enthesitis-related JIA, psoriatic arthritis, and undefined arthritis.

The pathophysiology mechanisms associated to JIA development are related to an abnormal activation of immune system cells such as B cells, T cells, natural killer (NK) cells, dendritic cells (DCs), monocytes, neutrophils, plasma cells, and to the production and release of pro-inflammatory mediators that ultimately lead to cartilage and bone destruction and systemic manifestations.

JIA has been classically considered a T-cell driven autoimmune disease, except for sJIA subtype, in which innate immune cells have a central role in disease pathogenesis. However, the detection of autoantibodies reacting with different target antigens in JIA patients suggests a central role of B cells in JIA pathophysiology.

Therapeutic intervention of jia begins at diagnosis with non-steroidal anti-inflammatory drugs (NSAIDs) followed by disease-modifying anti-rheumatic drugs (DMARDs, most often methotrexate) and/or corticosteroid intra-articular injection.

NSAIDs obtain both analgesic and anti-inflammatory effects. Local corticosteroid joint injections are effective in synovitis and may be a first-line treatment for oligoarthritis alone or in addition to DMARDs. Systemic administration of high dose corticosteroids provides good short-term effect, especially in sJIA patients.

The American College of Rheumatology (ACR) recommends early use of DMARDs, specifically MTX, leflunomide and/or sulfasalazine.

MTX is considered to be the first choice DMARD for oligo- and pJIA when NSAIDs and intraarticular steroids are insufficient.

MTX is also considered to be effective in children with PsJIA, though the axial manifestations limits prescription of MTX and so TNF inhibitors are typically required in these cases.

Leflunomide may be used as an alternative DMARD for pJIA in cases of MTX intolerance.

Sulfasalazine is recommended for patients with moderate activity of ERA with active peripheral arthritis, but is inefficient in case of sacroiliitis.

The emergence of biologic treatments has changed the prognosis for many JIA patients, whose condition did not improve adequately on conventional synthetic disease modifying anti-rheumatic drugs (csDMARDs), mainly methotrexate, or experienced side effects because of them. TNF-α inhibitors, such as etanercept, adalimumab , infliximab are widely used in JIA. In fact, etanercept is one of the most frequently prescribed biologics for JIA in many countries, including the United Kingdom. (19) Other biologics include tocilizumab , anakinra and canakinumab , abatacept and rituximab . The efficacy of biologics varies depending on the disease subtype.

Most healthy children have episodes of mild infections during the first years of life. In most cases, these episodes are respiratory or gastrointestinal viral infections. Children with juvenile idiopathic arthritis (JIA) have an allegedly higher risk of infection compared with healthy children because of their underlying condition.

Treatments used in JIA include corticosteroids, disease-modifying antirheumatic drugs (DMARDs), and biologic agents, all of which can increase the frequency of common mild infections and the risk of severe and opportunistic infections.

Disease-modifying anti-rheumatic drugs (DMARDs) help manage JIA by reducing inflammation and preventing joint damage, slowing the progression of the disease.

These therapies work by suppressing the immune system, which can lead to infection, despite growing evidence regarding the efficacy and safety of these drugs for children with JIA, it is unclear whether these agents increase the risk of infections - or whether the risk is increased to all or to only specific infections.

Moreover, there is a proportional relationship between the severity of the disease and the intensity of the treatment administered, and this association might constitute a confounding factor when assessing susceptibility to infections.

Besides novel findings, there is still little data available regarding the alteration of immune cells which control infection.

ELIGIBILITY:
Inclusion Criteria:

* 1. Patient age is above 16 years old 2. Patients who classified JIA according to International League of Associations for Rheumatology ILAR criteria received DMARDS therapy and in inactive state of disease

Exclusion Criteria:

* 1. Patients with active JIA 2. Any patient with any autoimmune disease other than JIA 3. Acquired and congenital lymphopenia

Ages: 6 Months to 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: -1. Patient age is above 16 years old 2. Patients who classified JIA according to International League of Associations for Rheumatology ILAR criteria received DMARDS therapy and in inactive state of disease
Sampling Method: Probability Sample
Enrollment: 75 (Estimated)
Dates: Start 2024-07-15 (Estimated); Primary Completion 2025-06-15 (Estimated); Study Completion 2026-11-30 (Estimated)

PRIMARY OUTCOMES:
lymphopenia | 1 year
  lymphopenia in JIA patients receiving MTX and biological therapy

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Oliveira-Ramos F, Eusebio M, M Martins F, Mourao AF, Furtado C, Campanilho-Marques R, Cordeiro I, Ferreira J, Cerqueira M, Figueira R, Brito I, Canhao H, Santos MJ, Melo-Gomes JA, Fonseca JE. Juvenile idiopathic arthritis in adulthood: fulfilment of classification criteria for adult rheumatic diseases, long-term outcomes and predictors of inactive disease, functional status and damage. RMD Open. 2016 Sep 22;2(2):e000304. doi: 10.1136/rmdopen-2016-000304. eCollection 2016. PMID 27752356
- [Background] Oliveira Ramos F, Rodrigues A, Magalhaes Martins F, Melo AT, Aguiar F, Brites L, Azevedo S, Duarte AC, Furtado C, Mourao AF, Sequeira G, Cunha I, Figueira R, Melo Gomes JA, Santos MJ, Fonseca JE. Health-related quality of life and disability in adults with juvenile idiopathic arthritis: comparison with adult-onset rheumatic diseases. RMD Open. 2021 Nov;7(3):e001766. doi: 10.1136/rmdopen-2021-001766. PMID 34819385
- [Background] Petty RE, Southwood TR, Manners P, Baum J, Glass DN, Goldenberg J, He X, Maldonado-Cocco J, Orozco-Alcala J, Prieur AM, Suarez-Almazor ME, Woo P; International League of Associations for Rheumatology. International League of Associations for Rheumatology classification of juvenile idiopathic arthritis: second revision, Edmonton, 2001. J Rheumatol. 2004 Feb;31(2):390-2. No abstract available. PMID 14760812
- [Background] Zaripova LN, Midgley A, Christmas SE, Beresford MW, Baildam EM, Oldershaw RA. Juvenile idiopathic arthritis: from aetiopathogenesis to therapeutic approaches. Pediatr Rheumatol Online J. 2021 Aug 23;19(1):135. doi: 10.1186/s12969-021-00629-8. PMID 34425842